CLINICAL TRIAL: NCT01405989
Title: An Open-label, Randomized, Two-period Crossover Study to Evaluate the Effect of Multiple Doses of Ketoconazole on the Pharmacokinetics of Darexaban and Metabolites in Young Healthy Male Subjects
Brief Title: To Evaluate if Multiple Doses of Ketoconazole Change the Blood Concentration of YM150 (Darexaban)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150-CL-037; 2009-015761-32 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2011-07

CONDITIONS: Pharmacokinetics of Darexaban and Metabolites; Healthy Subjects
Keywords: Pharmacokinetics; darexaban; ketoconazole; Phase 1
MeSH Terms: interventions — darexaban; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm A (Experimental): darexaban, wash-out, ketoconazole + darexaban
  Interventions: Drug: darexaban; Drug: ketoconazole
- Treatment arm B (Experimental): ketoconazole + darexaban, wash-out, darexaban
  Interventions: Drug: darexaban; Drug: ketoconazole

INTERVENTIONS:
Drug: darexaban — oral
  Other Names: YM150
Drug: ketoconazole — oral
  Other Names: Nizoral

SUMMARY:
The primary objective of this study is to determine the effect of ketoconazole on the blood concentrations of darexaban and its metabolites (drug degradation products). The secondary objective of the study is to evaluate the safety and tolerability of a single dose of darexaban alone and when administered together with ketoconazole.

DETAILED DESCRIPTION:
This is an open-label, 2-period crossover study in young healthy male subjects to evaluate the effect of multiple once daily doses of ketoconazole on the pharmacokinetics (PK) of darexaban and metabolites after a single dose of darexaban. In addition, safety and tolerability of darexaban administered alone and in combination with ketoconazole, is evaluated. Eligible subjects are admitted to the clinical unit in the morning of Day -1. The subjects are randomized to receive either first darexaban plus ketaconazole and then darexaban alone, or first darexaban alone followed by darexaban plus ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5-30.0 kg/m2
* Male subjects must be non-fertile, i.e. surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies

Exclusion Criteria:

* Known or suspected hypersensitivity to darexaban or ketoconazole or any components of the formulation used
* Any of the liver function tests (i.e. ALT, AST and bilirubin) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units (210 g) of alcohol per week within the 3 months prior to study
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of darexaban and its metabolites assessed by plasma concentration | Plasma samples are taken until 72 hours (darexaban alone) or 144 hours (combination of darexaban and ketoconazole) after darexaban dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — SGS Aster, Paris, France
Locations (1):
- SGS Aster, Paris, France